CLINICAL TRIAL: NCT00752375
Title: A Randomized Controlled Trial of Antibiotic Prophylaxis in Children With Pyelonephritis in the Abscence of Vesicoureteral Reflux
Brief Title: Antibiotic Prophylaxis in Children With Pyelonephritis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No participants
Sponsor: University of Alberta (Other)
Collaborators: Canadian Urological Association (Industry)
Responsible Party: Principal Investigator, Darcie Kiddoo, Physician, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6545
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Pyelonephritis
Keywords: pyelonephritis; pediatric pyelonephritis; vesicoureteral reflux; DMSA scan
MeSH Terms: conditions — Pyelonephritis; Vesico-Ureteral Reflux | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; bacitracin zinc, neomycin sulfate, polymyxin B, drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Eligible children will be randomized to antibiotic prophylaxis. Children under 3 months will receive amoxicillin 10mg/kg once per day. Children >3months will receive Trimethoprim Sulfamethoxazole (2mg/kg Trimethoprim component). Those children with a Sulfa allergy will receive nitrofurantoin (1mg/kg) once per day.
  Interventions: Drug: Trimethoprim Sulfamethoxazole
- B (Placebo Comparator): Eligible children will then be randomized to placebo.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Trimethoprim Sulfamethoxazole — * Children >3months of age will receive Trimethoprim Sulfamethoxazole (2mg/kg Trimethoprim component)per day for one year.
  * Children under 3 months of age will receive amoxicillin 10mg/kg once per day for one year.
  * Those children with a Sulfa allergy will receive nitrofurantoin (1mg/kg) once per day for one year.
  Other Names: Septa; Bactrim
  Arms: A
Drug: placebo — * Placebo matching Trimethoprim Sulfamethoxazole (2mg/kg Trimethoprim component)for children more than 3 months of age
  * Placebo matching amoxicillin 10mg/kg once per day for children under 3 months of age
  * Placebo matching nitrofurantoin (1mg/kg) once per day for children with a sulfa allergy.
  Arms: B

SUMMARY:
Children who present with pyelonephritis undergo many investigations, and long term care to prevent renal damage. The focus is primarily on preventing renal failure however along the way and particularly with children, other issues arise which impact their lives, as well as their family's lives. Parents are concerned about subjecting their children to invasive procedures and long term antibiotic use, particularly if they are not sure of the benefit. This study seeks to provide information on the impact of investigation and long term antibiotic treatment in reference to long term health and quality of life in children who present with febrile urinary tract infections in the absence of anatomic abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Children 0 to 12 years of age presenting with first episode of acute pyelonephritis in the absence of vesicoureteral reflux.
* Acute pyelonephritis defined as presence of fever, a positive urine culture (growth of a single urinary tract pathogen at =10(8) CFU/ml for catheterization specimens and =10(4) CFU/ml for clean catch specimens), and a positive DMSA scan (a discreet defect or generalized decrease in activity).

Exclusion Criteria:

* Neurogenic bladder
* anatomic congenital anomaly
* allergy to all prophylactic antibiotics
* children whose parents do not wish to participate

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To determine whether antibiotic prophylaxis prevents recurrent urinary tract infections by assessing if there is a decreased incidence of urinary tract infections. | one year

SECONDARY OUTCOMES:
To determine whether antibiotic prophylaxis prevents long-term renal scarring by assessing results of DMSA scans to look at long term renal scarring. | One year and five years
To determine whether recurrent infections and involvement with the medical system impacts quality of life by assessing how this medical condition affects children using standardized quality of life questionnaires. | Yearly for five years

CONTACTS AND LOCATIONS:
Overall Officials: Darcie Kiddoo, MD, Principal Investigator — University of Alberta
Locations (1):
- Stollery Children's Hospital, Edmonton, Alberta, Canada